CLINICAL TRIAL: NCT07178964
Title: THE USE OF POTASSIUM-RICH SALT SUBSTITUTES IN BLOOD PRESSURE CONTROL OF KIDNEY TRANSPLANT RECIPIENTS
Brief Title: POTASSIUM-RICH SALT SUBSTITUTES IN KIDNEY TRANSPLANT RECIPIENTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tanja Belčič Mikič, MD, PhD, FEBTM, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250138
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension Arterial; Kidney Transplant
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium-enriched salt-substitute arm (Experimental): The patients in this arm will use potassium-enriched salt-substitutes for cooking and seasoning food in their home environment.
  Interventions: Other: Potassium-enriched salt-substitute
- Regular table salt arm (Sham Comparator): The patients in this arm will use regular table salt for cooking and seasoning food in their home environment.
  Interventions: Other: Regular table salt

INTERVENTIONS:
Other: Potassium-enriched salt-substitute — The patients in the experimental group will use potassium-enriched salt-substitutes for cooking and seasoning food in their home environment. Potassium-enriched salt-substitutes will contain 25% potassium chloride nad 75% sodium chloride.
  Arms: Potassium-enriched salt-substitute arm
Other: Regular table salt — Patients in this arm will use regular table salt (100 % sodium chloride) for cooking and seasoning food in their home environment.
  Arms: Regular table salt arm

SUMMARY:
Excessive sodium intake and inadequate potassium intake in the diet are known risk factors for the development of arterial hypertension and an increased risk of cardiovascular events. Data from randomized controlled trials show that the use of salt substitutes with reduced sodium and increased potassium content represent an effective way to reduce dietary sodium intake, blood pressure and the occurrence of cardiovascular events. Patients adhere well to the use of salt substitutes as they do not have to change their daily cooking and seasoning habits and the taste is comparable to that of regular salt. The World Health Organization (WHO) also suggests the use of salt substitutes as an acceptable strategy for reducing dietary salt intake and thus lowering blood pressure and the burden of cardiovascular disease. Recommendations for the use of salt substitutes are not uniform, primarily because of the potential risk of adverse events with increased potassium intake in some individuals, such as patients with advanced chronic kidney disease (CKD), patients receiving potassium-sparing diuretics, and patients receiving potassium supplements.

Nephrology guidelines rarely comment on the use of potassium-rich salt substitutes or discourage their use in patients with advanced stage 4 and 5 CKD, with the exception of Chinese guidelines, which mention the use of potassium-rich salt substitutes in CKD patients not on dialysis depending on serum potassium levels. CKD patients have largely been excluded from clinical trials of potassium-rich salt substitutes, so there is insufficient data on their safety and efficacy in CKD patients.

In this randomized controlled trial, we will investigate the effects of using potassium-enriched salt substitutes on blood pressure control and serum potassium levels in kidney transplant recipients. In the intervention group, patients will use potassium-enriched salt substitutes at home in a ratio of 75% sodium chloride and 25% potassium chloride instead of regular table salt (100% sodium chloride) for cooking and seasoning food. In the control group, patients will use regular salt at home for cooking and seasoning food. The intervention and control groups will each include 40 to 50 patients who will be monitored for 12 weeks. The study's main focus will be the change in serum potassium and blood pressure before and after the intervention.

We expect to confirm the positive effects of potassium-enriched salt substitutes on blood pressure in kidney transplant recipients without causing undesirable hyperkalemia.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality worldwide, especially in patients with chronic kidney disease and kidney transplantation. Arterial hypertension is one of the most important risk factors for the occurrence of cardiovascular diseases. Despite advances in modern medicine, the treatment of arterial hypertension is often a major challenge, partly due to patients' poor adherence to medication and lifestyle changes, including adherence to dietary recommendations.

In addition to a reduced sodium intake, an increased potassium intake also plays an important role in lowering blood pressure. The mechanism of increased sodium intake in the development of high blood pressure is probably related to the inability of the kidneys to excrete excess sodium. Potassium deficiency leads to additional sodium retention as it stimulates the activation of the sympathetic nervous system and the renin-angiotensin-aldosterone system. Conversely, an increased potassium intake has the effect of reducing salt sensitivity. Increased potassium intake inhibits the phosphorylation of the NaCl cotransporter and simultaneously reduces sodium reabsorption in the proximal tubule and/or in the ascending limb of the loop of Henle.

Numerous epidemiological studies have shown an inverse relationship between potassium intake and blood pressure. The large international INTERSALT study showed that systolic blood pressure falls by an average of 2 to 3 mmHg when potassium intake is increased by 30 to 45 mmol/day. Reducing sodium intake and increasing potassium intake is likely to be an effective measure for treating arterial hypertension and cardiovascular disease in the population.

Recommendations for the use of salt substitutes to lower blood pressure and prevent cardiovascular disease are not uniform, primarily because of the potential risk of adverse events (especially hyperkalemia) with increased potassium intake in certain individuals such as patients with advanced chronic kidney disease (CKD), patients receiving potassium-sparing diuretics and patients receiving potassium supplements.

Nephrology guidelines rarely mention the use of potassium-rich salt substitutes or advise against it in patients with advanced CKD stages 4 and 5, with the exception of Chinese guidelines, which mention the use of potassium-enriched salt substitutes in non-dialysis CKD patients, depending on the serum potassium level. CKD patients have been mostly excluded from clinical studies of the use of potassium-enriched salt substitutes, so there is not enough data available for CKD patients on the safety and efficacy of potassium-enriched salt substitutes.

A review of the literature suggests that different sources of potassium (diet or potassium supplements) have different effects on serum potassium levels in patients with CKD. The effect of potassium-enriched salt substitutes on serum potassium levels in renal patients is unknown. A study is currently underway in the United States to study the effect of salt substitutes on serum potassium and blood pressure in hemodialysis patients. Since this is a population of patients at increased risk for hyperkalemia, the primary goal is safety, namely the detection of hyperkalemia.

In this randomized single-blind controlled trial, we want to examine the effect of using potassium-enriched salt substitutes on serum potassium and blood pressure in kidney transplant patients with hypertension. In the intervention group, patients will use potassium-enriched salt substitutes at home in a ratio of 75% sodium chloride and 25% potassium chloride instead of regular table salt for cooking and seasoning food. In the control group, patients will use table salt (100% sodium chloride) at home for cooking and seasoning food. Potassium-enriched salt substitutes and 100% sodium chloride will be prepared for patients in the hospital pharmacy. During the study, we will not introduce new antihypertensive medications or medications that affect serum potassium. If the patient is receiving potassium supplements before inclusion in the study, they will be discontinued at least a week before the start of the study. Before the start of the intervention, we will measure the patients' body composition and check the patients' dietary habits using a questionnaire. After the intervention, the patients will report any changes in the taste of home-cooked food.

The main purpose of the study is:

* to show that the use of salt substitutes in kidney transplant patients does not lead to a significantly increased risk of hyperkalemia.
* to show that the use of salt substitutes in kidney transplant recipients has an effect on lowering blood pressure and is thus a safe and effective measure in the management of arterial hypertension in this population.

We expect a mild effect on blood pressure reduction in kidney transplant recipients with no significant increased risk of hyperkalemia.

ELIGIBILITY:
Inclusion Criteria:

* patients with a transplanted kidney ≥ 3 months post kidney-transplant
* a functioning transplanted kidney with estimated glomerular filtration rate (eGFR) according to CKD/EPI equation of at least 25 ml/min
* Elevated blood pressure/hypertension at the time of examination at the Kidney Transplantation Center outpatient clinic, determined by standardized blood pressure measurement (RR ≥ 130/80 mmHg)
* Age ≥ 18 years

Exclusion Criteria:

* eGFR according to CKD/EPI equation below 25 ml/min
* serum potassium > 5 mmol/l
* history of unexplained hyperkalemia
* pregnancy or planning of pregnancy
* inability to provide informed consent or to participate in the study (mental retardation, psychiatric illness in an uncontrolled phase)
* multiple organ transplantation
* Consuming most of daily meals outside the home environment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hyperkalemia | 12 weeks.
  Change in serum potassium in mmol/l after using potassium-enriched salt-substitutes for cooking and seasoning food at home for 12 weeks

SECONDARY OUTCOMES:
Change in systolic blood pressure | 12 weeks
  Change in systolic blood pressure in mmHg measured with standardized office blood-pressure measurement
Change in diastolic blood pressure | 12 weeks
  Change in diastolic blood pressure in mmHg measured with standardized office blood pressure measurement
Change in average systolic 24-hour blood pressure | 12 weeks
  Change in average 24-hour systolic blood pressure measured by 24-hour blood pressure monitoring device
Change in average diastolic 24-hour blood pressure | 12 weeks
  Change in average 24-hour diastolic blood pressure measured by 24-hour blood pressure monitoring device
Change in average daily systolic blood pressure | 12 weeks
  Change in average daily systolic blood pressure measured by 24-hour blood pressure monitoring device
Change in average daily diastolic blood pressure | 12 weeks
  Change in average daily diastolic blood pressure measured by 24-hour blood pressure monitoring device
Change in average night systolic blood pressure | 12 weeks
  Change in average night systolic blood pressure measured by 24-hour blood pressure monitoring device
Change in average night diastolic blood pressure | 12 weeks
  Change in average diastolic night blood pressure measured by 24-hour blood pressure measuring device
Reduction in the number or dose of antihypertensive drugs | 12 weeks
  A reduction in the number or dose of used antihypertensive drugs to achieve target blood pressure
Change in the urine sodium/potassium ratio | 12 weeks
  Change in the ratio of sodium to potassium excreted in urine, based on measurements of 24-hour urine collection
Change in taste of food | 12 weeks
  Patients will report on change of the taste of food (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Belcic Mikic, MD, PhD, FEBTM, Principal Investigator — University Medical Centre Ljubljana; Miha Arnol, Professor, MD, PhD, FEBTM, Study Director — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request from the principal investigator in an anonymized form.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 30.09.2026-30.09.2027

REFERENCES:
- [Background] Chia YC, He FJ, Cheng MH, Shin J, Cheng HM, Sukonthasarn A, Wang TD, Van Huynh M, Buranakitjaroen P, Sison J, Siddique S, Turana Y, Verma N, Tay JC, Schlaich MP, Wang JG, Kario K; HOPE-Asia Network. Role of dietary potassium and salt substitution in the prevention and management of hypertension. Hypertens Res. 2025 Jan;48(1):301-313. doi: 10.1038/s41440-024-01862-w. Epub 2024 Oct 29. PMID 39472546
- [Background] Romero-Gonzalez G, Rodriguez-Chitiva N, Canameras C, Paul-Martinez J, Urrutia-Jou M, Troya M, Soler-Majoral J, Graterol Torres F, Sanchez-Baya M, Calabia J, Bover J. Albuminuria, Forgotten No More: Underlining the Emerging Role in CardioRenal Crosstalk. J Clin Med. 2024 Jan 29;13(3):777. doi: 10.3390/jcm13030777. PMID 38337471
- [Background] Xu X, Zeng L, Jha V, Cobb LK, Shibuya K, Appel LJ, Neal B, Schutte AE. Potassium-Enriched Salt Substitutes: A Review of Recommendations in Clinical Management Guidelines. Hypertension. 2024 Mar;81(3):400-414. doi: 10.1161/HYPERTENSIONAHA.123.21343. Epub 2024 Jan 29. PMID 38284271
- [Background] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- [Background] Visser WJ, Gritter M, Hoorn EJ. Dietary Potassium in Chronic Kidney Disease: Do Not Restrict the Evidence. J Ren Nutr. 2021 Nov;31(6):552-553. doi: 10.1053/j.jrn.2020.12.012. Epub 2021 Mar 12. No abstract available. PMID 33715954
- [Background] Daneshzad E, Hatami SE, Sobhani S, Ghoreshi B, Khonsari NM, Shahrestanaki E, Pezeshki M, Kiaee ZF, Assar O, Qorbani M. Effects of potassium-enriched salt substitutes on blood pressure in Iranian hypertensive patients: the protocol for a randomised, double-blind controlled trial. BMJ Open. 2025 Jun 25;15(6):e090472. doi: 10.1136/bmjopen-2024-090472. PMID 40562554
- [Background] Tsai YC, Tsao YP, Huang CJ, Tai YH, Su YC, Chiang CE, Sung SH, Chen CH, Cheng HM. Effectiveness of salt substitute on cardiovascular outcomes: A systematic review and meta-analysis. J Clin Hypertens (Greenwich). 2022 Sep;24(9):1147-1160. doi: 10.1111/jch.14562. PMID 36196475
- [Background] Bernabe-Ortiz A, Sal Y Rosas VG, Ponce-Lucero V, Cardenas MK, Carrillo-Larco RM, Diez-Canseco F, Pesantes MA, Sacksteder KA, Gilman RH, Miranda JJ. Effect of salt substitution on community-wide blood pressure and hypertension incidence. Nat Med. 2020 Mar;26(3):374-378. doi: 10.1038/s41591-020-0754-2. Epub 2020 Feb 17. PMID 32066973
- [Background] Eleftheriadis G, Naik MG, Osmanodja B, Halleck F, Schrezenmeier E, Liefeldt L, Choi M, Bachmann F, Avaniadi DP, von Hoerschelmann E, Lucht C, Zaks M, Duettmann W, Budde K. Office or home versus 24-h blood pressure measurement in stable kidney transplant recipients. Nephrol Dial Transplant. 2024 Oct 30;39(11):1890-1899. doi: 10.1093/ndt/gfae076. PMID 38549427
- [Background] Tantisattamo E, Molnar MZ, Ho BT, Reddy UG, Dafoe DC, Ichii H, Ferrey AJ, Hanna RM, Kalantar-Zadeh K, Amin A. Approach and Management of Hypertension After Kidney Transplantation. Front Med (Lausanne). 2020 Jun 16;7:229. doi: 10.3389/fmed.2020.00229. eCollection 2020. PMID 32613001
- [Background] Speer C, Benning L, Morath C, Zeier M, Frey N, Opelz G, Dohler B, Tran TH; Collaborative Transplant Study. Blood Pressure Goals and Outcomes in Kidney Transplant Recipients in an Analysis of the Collaborative Transplant Study. Kidney Int Rep. 2024 Dec 6;10(3):780-790. doi: 10.1016/j.ekir.2024.12.004. eCollection 2025 Mar. PMID 40225383